CLINICAL TRIAL: NCT04755296
Title: Response of Aerobic Capacity to Low Level Laser Therapy in Burned Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Noha Mohamed Kamel, lecturer at Department of Physical Therapy for Surgery, Faculty of Physical Therapy, Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Aerobic capacity in burns
Record Dates: First submitted 2021-02-06; First posted 2021-02-16 (Actual); Last update posted 2021-02-16 (Actual); Status verified 2021-02

CONDITIONS: Burns
MeSH Terms: conditions — Burns | interventions — Low-Level Light Therapy; Exercise

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low level laser therapy and aerobic exercises group (Experimental): They received low level laser therapy and aerobic exercises using a treadmill, 3 sessions per week for 12 weeks.In addition to traditional physical therapy program in the form of (stretching and strengthening exercises for all affected areas, diaphragmatic breathing exercises and activities of daily living).
  Interventions: Device: Low level laser therapy; Other: Aerobic exercises; Other: Traditional physical therapy program
- Control group (aerobic exercises group) (Active Comparator): They received aerobic exercises 3 times weekly for 12 weeks.In addition to the same traditional physical therapy program.
  Interventions: Other: Aerobic exercises; Other: Traditional physical therapy program

INTERVENTIONS:
Device: Low level laser therapy — Low level laser therapy was applied immediately before each aerobic exercise training session by using a multidiode cluster (with four diode spots; Polaris2, manufactured by Astar ABR, Poland) )on 12 sites on the lower limb (6 on quadriceps ( 2 centrally on rectus femoris and vastus intermedius,2 laterally on vastus lateralis, and two medially on vastus medialis), 4 on hamstrings and 2 on gastrocnemius) with the following parameters: 808 nm, continous output, 200 mW each diode (total of 800 mW) power output, 24 J energy on each site (6 J for each spot) , 40 seconds at each site (8 minutes of total treatment time in lower limb) and 288 J total energy delivered per lower limb, 48 irradiation points per lower limb ,3 sessions weekly for 12 weeks.
  Arms: Low level laser therapy and aerobic exercises group
Other: Aerobic exercises — Aerobic exercise program consisted of walking on the treadmill at a rate of 3 sessions/week for 12 weeks, with each session lasting for 40 minutes in the form of warming up for 5 minutes at intensity of <50% of the previously determined VO2max of each participant, 30 minutes of treadmill exercises at intensity of (70-85%) of the previously determined VO2max of each participant then 5 minutes cooling down at intensity of<50% of the previously determined VO2max of each participant.
Other: Traditional physical therapy program — Patients were received traditional physical therapy program in the form of (stretching and strengthening exercises for all affected areas, diaphragmatic breathing exercises and activities of daily living).

SUMMARY:
Severe burns can decrease pulmonary function and impair aerobic capacity persisting for long times post injury. Low level laser therapy is a new modality used to improve aerobic capacity, enhance exercise performance, increase time until fatigue when used prior to aerobic exercises. This study aimed to evaluate the effects of pre- exercise low level laser therapy on aerobic capacity in burned patients.

DETAILED DESCRIPTION:
Low level laser therapy has a beneficial therapeutic effect on promoting aerobic capacity, improving maximum oxygen consumption and increasing treadmill time when preceding aerobic exercise training.This study was conducted to determine the effects of pre- exercise low level laser therapy on aerobic capacity in burned patients. Low level laser therapy was applied to the study group for 12 weeks before aerobic exercises, three sessions / week, while control group received 12 weeks of aerobic exercises, three times weekly. Patients in both groups were received the traditional physical therapy program as a routine treatment. Aerobic capacity was assessed by measuring maximum oxygen consumption and time to exhaustion at baseline and after twelve weeks of interventions for both groups.

ELIGIBILITY:
Inclusion Criteria:

* Sixty adult burned patients were selected under the following criteria:

  * Patients were both males and females.
  * Their age ranged from (25-40) years.
  * Patients suffered from second degree thermal burns with total body surface area(TBSA) for burns ranged from 20-40%.
  * Patients were participated in this study one month after their hospital discharge.

Exclusion Criteria:

* Cardiopulmonary diseases.
* Any limitation in range of motion (ROM) of joints of the lower limbs which may prevent adequate participation in aerobic exercise program.
* Leg amputation.
* Quadriplegia.
* Psychological illness or severe behavior or cognitive disorders.
* Patients who participated in any rehabilitation program before the study that may affect the results of the study.

Ages: 25 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Aerobic capacity was assessed by measuring maximum oxygen consumption (VO2max) | 12 weeks
  Aerobic capacity was evaluated by measuring VO2max during a Graded Exercise Test (GXT) performed on a treadmill using the modified Bruce protocol before the treatment and after 12 weeks of treatment for both groups.The Bruce protocol required subjects to walk at progressively higher workloads, with the treadmill speed and the inclination were increased incrementally every 3 minutes until it was no longer possible for the participant to continue. During GXT, participants breathed through a face mask which was linked to a calibrated expired gas analysis system (UltimaTM Series, Cardiorespiratory Diagnostic systems),MED GRAPHICSTM, St. Paul, Minnesota ,USA. Expired gas passed through a flowmeter, oxygen and carbon dioxide analyzers which were connected to a computer, which measured oxygen uptake.The sum of the 4 highest successive 15 s VO2 values was recorded as VO2max of the participants.

SECONDARY OUTCOMES:
Time to exhaustion (Treadmill time) | 12 weeks
  Time to exhaustion (Treadmill time) was measured by calculating the maximum time that the patient could walk on the treadmill.

CONTACTS AND LOCATIONS:
Overall Officials: N M Kamel, PhD, Principal Investigator — Cairo University
Locations (1):
- Cairo University, Cairo, Egypt

REFERENCES:
- [Background] Grisbrook TL, Wallman KE, Elliott CM, Wood FM, Edgar DW, Reid SL. The effect of exercise training on pulmonary function and aerobic capacity in adults with burn. Burns. 2012 Jun;38(4):607-13. doi: 10.1016/j.burns.2011.11.004. Epub 2012 Feb 16. PMID 22342175
- [Background] De Marchi T, Leal Junior EC, Bortoli C, Tomazoni SS, Lopes-Martins RA, Salvador M. Low-level laser therapy (LLLT) in human progressive-intensity running: effects on exercise performance, skeletal muscle status, and oxidative stress. Lasers Med Sci. 2012 Jan;27(1):231-6. doi: 10.1007/s10103-011-0955-5. Epub 2011 Jul 8. PMID 21739259
- [Background] Miranda EF, Tomazoni SS, de Paiva PRV, Pinto HD, Smith D, Santos LA, de Tarso Camillo de Carvalho P, Leal-Junior ECP. When is the best moment to apply photobiomodulation therapy (PBMT) when associated to a treadmill endurance-training program? A randomized, triple-blinded, placebo-controlled clinical trial. Lasers Med Sci. 2018 May;33(4):719-727. doi: 10.1007/s10103-017-2396-2. Epub 2017 Nov 29. PMID 29185134